CLINICAL TRIAL: NCT06651970
Title: A Multicentre, Open-label, Randomised Phase IV Study to Investigate Acalabrutinib Monotherapy Compared to Investigator's Choice of Treatment in Adults (> 18 Years) With Chronic Lymphocytic Leukaemia and Moderate to Severe Cardiac Impairment
Brief Title: Acalabrutinib Monotherapy vs Investigator's Choice of Treatment in Patients With CL Leukaemia and Heart Failure
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Fortrea (Industry); CALYX Inc. (Unknown); eResearch Technology, Inc. (Industry); CISCRP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D8223C00016
Record Dates: First submitted 2024-08-20; First posted 2024-10-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukaemia; Heart Failure
Keywords: Hemic Diseases; Lymphatic Diseases
MeSH Terms: conditions — Leukemia, B-Cell; Heart Failure; Lymphatic Diseases | interventions — acalabrutinib; Rituximab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Acalabrutinib Monotherapy) (Active Comparator): All participants randomised to Arm A will receive treatment with the investigational product acalabrutinib.
  Interventions: Drug: Acalabrutinib
- Treatment Arm B (Other): Patients in Arm B will receive investigator's choice of treatment its duration will be based on standard duration of therapy for that regimen or until disease progression/patient withdrawal/study termination, whichever occurs first.
  Interventions: Other: Investigator's choice of treatment

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib Monotherapy
  Other Names: Calquence
  Arms: Treatment Arm A (Acalabrutinib Monotherapy)
Other: Investigator's choice of treatment — control arm treatment type will be defined by the PI prior to randomisation
  Other Names: Investigator's choice of treatment : i.e venetoclax, Rituximab, Obinutuzumab, Zanubrutinib etc.
  Arms: Treatment Arm B

SUMMARY:
This will be a global Phase IV, open-label, randomised study to evaluate the safety and tolerability of acalabrutinib (monotherapy, 100 mg orally [po], twice daily [bd]) compared to investigator's choice of treatment, in patients with CLL (TN or R/R) and moderate to severe cardiac impairment. All patients will have cardiac impairment as defined by LVEF of < 50%.

Randomisation will be stratified by LVEF > 40% vs ≤ 40% to stratify for moderate and severe cardiac impairment, which for this study are defined as follows:

Severe cardiac impairment: in those with LVEF ≤ 40% Moderate cardiac impairment: in those with LVEF > 40% to < 50%. The study is planned to take place in approximately 20 centres globally. The study will be conducted in centres that have established close collaboration between the Haematology and Cardiology divisions, preferably with a cardio-oncologist on the team.

An IDMC will be responsible for making recommendations for study continuation.

DETAILED DESCRIPTION:
Randomised controlled study:

Treatment phase:

Patients will receive treatment with either acalabrutinib 100 mg po tablets bd (until unacceptable toxicity or progression) or investigator's choice of treatment (chlorambucil, venetoclax, ibrutinib, zanabrutinib, rituximab or Obinutuzumab etc). For the control arm the treatment type and duration will be defined by the PI prior to randomisation.

Each treatment cycle is 28 days/4 weeks. Haematology visits (labs, physical exam), will be performed at the first day of each cycle for the first 8 cycles and every 4 cycles there after.

Response assessment will be performed by the PI in accordance with modified iwCLL 2018 criteria every 4 cycles (16 weeks). Imaging and BM testing only as deemed appropriate by PI.

Safety assessments will be performed at every visit.

Cardiology assessments will be performed at the end of cycle 1 (C2D1) and 3 (C4D1) and thereafter every 4 cycles (16 weeks). These assessments will include:

* A cardiology consult.
* ECHO, 12-lead ECG and 24-hour Holter.
* Cardiac biomarkers.
* Any additional testing will be performed as clinically indicated.

Cardiac MRI post-screening will be performed every year.

Decisions for permanent withdrawal or modifications to treatment due to cardiac AEs will be made by PI after close consultation with the cardiologist.

Post-Treatment Phase:

Safety assessments

Once treatment is discontinued due to any of the reasons mentioned above, a safety follow-up (SFU) will occur within 45 days of the last dose of treatment. This will occur regardless of the patient developing progressive disease or initiation a new anti-CLL therapy during that timespan. The evaluation will include:

* Cardiology consult
* Cardiac biomarkers
* 12-lead ECG, ECHO and 24 hour Holter
* Cardiac MRI (if not performed in the last 6 months).

The subsequent safety assessments will continue until disease progression, WoC, death or termination of study whichever occurs first.

These will mirror the in-treatment schedule, with cardiology consults including ECHO, ECG, cardiac biomarkers and 24 hour Holter performed every 16 weeks and yearly cardiac MRI. Once patient has progressive disease they will be contacted to assess survival status every 16 weeks.

Response assessments Patients that discontinue treatment prior to progression will continue to be evaluated for disease progression every 16 weeks. The response assessment will be per iwCLL 2018 guidelines and will be performed by the PI. Bone marrow testing and imaging will continue to remain optional and per PI discretion.

Once patient has progressive disease they will be contacted every 16 weeks for survival status and information on any new anti-cancer therapy until WoC, death, termination of study by Sponsor whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age, at the time of signing the informed consent.
2. Eastern Cooperative Oncology Group performance status of 0 to 3
3. Left ventricular ejection fraction assessed by ECHO < 50%.
4. Diagnosis of CLL
5. Treatment naïve or relapsed/refractory patients who received no more than 2 prior lines of systemic anti-CLL treatment.
6. Active disease per iwCLL 2018 criteria that requires treatment.
7. Meet the following laboratory parameters:

   1. Absolute neutrophil count (ANC) ≥ 500 cells/μL (0.50 × 109/L).
   2. Platelet count ≥ 30,000 cells/μL (30 × 109/L).
   3. Serum aspartate aminotransferase and ALT ≤ 3.0 × ULN.
   4. Total bilirubin ≤ 1.5 × ULN unless directly attributable to Gilbert's syndrome.
   5. Estimated creatinine clearance (ie, estimated glomerular filtration rate [eGFR] using Cockcroft-Gault) ≥ 40 mL/min, or serum creatinine ≤ 2 × ULN.
8. Women and men who are sexually active and can bear children must agree to use highly effective forms of contraception while on the study and for 2 days after the last dose of acalabrutinib.
9. Patients must be willing and able to adhere to the study visit schedule, understand, and comply with other protocol requirements, and provide written informed consent and authorisation to use protected health information (in accordance with national and local patient privacy regulations). Note: vulnerable patients, as defined in the ICH GCP, are not allowed on this protocol (eg, prisoners or institutionalised patients).

Exclusion Criteria:

1. Known active CNS leukaemia, leptomeningeal disease or spinal cord compression. In case of R/R patients with prior history of CNS localisation of leukaemia who received treatment are eligible provided that there is no evidence of CNS involvement at study entry as documented by cerebrospinal fluid (CSF) cytology and/or brain MRI.
2. Ongoing Richter's transformation.
3. Prior exposure to a BTKi.
4. Major surgery within 30 days before first dose of study treatment.
5. Uncontrolled haemolytic anaemia.
6. Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study treatment.
7. Received a live virus vaccination within 28 days of first dose of study treatment.
8. History of or ongoing confirmed PML.
9. History of prior malignancy except for the following:

   1. Prior history of malignancy with no evidence of active disease present for more than

3 years before screening or felt to be at low risk for recurrence by treating physician.

(b) Adequately treated lentigo maligna melanoma without current evidence of disease or adequately resected non-melanomatous skin cancer (ie, basal cell carcinoma or squamous cell carcinoma of the skin). (c) Curatively treated in situ carcinoma of the cervix or carcinoma in situ of the prostate at any time prior to study without current evidence of disease. 10 Unable to swallow tablets or malabsorption syndrome, or disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or gastric bypass, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.

11 Active uncontrolled systemic infection (bacterial, fungal, viral or other) or clinically significant localised infection. 12 Known history of infection with human immunodeficiency virus (HIV). 13 Serologic status reflecting active HepB or HepC infection.

1. Patients with HepB core antibody positive who are surface antigen negative or who are HepC antibody positive will need to have a negative polymerase chain reaction (PCR) result before randomisation and must be willing to undergo deoxyribonucleic acid (DNA) PCR testing during the study.
2. Patients who are HepB surface antigen positive or HepB PCR positive and those who are HepC PCR positive will be excluded. 14 History of stroke or intracranial haemorrhage within 6 months prior to randomisation.

   15 History of bleeding diathesis (eg, haemophilia, von Willebrand disease). 16 Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days of first dose of study treatment. Direct anti-X (DOACs) or low molecular weight heparins (LMWH, eg, enoxaparin) on stable dosing schedule is allowed. 17 Requires treatment with a strong cytochrome P450 3A (CYP3A) inhibitor/inducer. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study treatment is prohibited. 18 Breastfeeding or pregnant. 19 Concurrent participation in another therapeutic clinical trial. 20 Uncontrolled cardiac/cardiovascular disease including the following:
   * Uncontrolled cardiac tachyarrhythmias (sinus, atrial or ventricular) that require new/additional therapy within the last month.
   * Clinically significant outlying QT interval corrected by Fridericia's formula (QTcF) values; QTcF > 470 ms or QTcF < 330 ms.
   * Unstable ischaemic heart disease (IHD), recent (< 3 months): episode of acute coronary syndrome, including acute myocardial infarction and unstable angina pectoris.
   * Percutaneous coronary intervention, or coronary artery bypass graft within the last month. 21 Uncontrolled hypertension despite optimal management. 22 Current life-threatening illness, medical conditions, organ system dysfunction or lifestyle habits which, in the investigator's opinion, could compromise the patient's safety or ability to adhere to the study protocol.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2030-08-16 (Estimated); Study Completion 2030-08-16 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints 1: To evaluate the incidence of CV (CardioVascular) adverse events leading to drug discontinuation after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Frequency and time to discontinuation of any study treatment due to worsening in cardiovascular function or cardiovascular AEs.
Safety endpoints 2: To evaluate the duration on treatment prior to drug discontinuation due to CV adverse events after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Incidence of Grade 4 and 5 cardiovascular events of interest.
Safety endpoints 3: To evaluate the incidence of life threatening and fatal cardiac events of interest after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Incidence and relationship to study treatment of Grade ≥ 3 AEs.
Safety endpoints 4: To evaluate the frequency of grade≥3 Adverse events after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Incidence and relationship to study treatment of Adverse events of special interest (AESI) defined per Acalabrutinib IB
Safety endpoints 5: To evaluate the frequency of AESI per Acalabrutinib IB after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Incidence and relationship to study treatment of Non-cardiovascular AE that led to discontinuation of any study treatment.
Safety endpoints 6: To evaluate the rate of discontinuation due to non-CV adverse events after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Incidence and relationship to study treatment of Events of clinical interest (ECI) per acalabrutinib IB
Safety endpoints 7: To evaluate the rate of any serious adverse event after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Incidence and relationship to study treatment of Serious adverse events (SAEs).

SECONDARY OUTCOMES:
Efficacy Endpoints 1:To evaluate the overall survival after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Overall survival (OS), defined as the time from randomisation to death from any cause.
  Per iwCLL 2018 criteria:
  • Event-free survival (EFS), defined as the time from randomisation to disease progression, initiation of subsequent anti-CLL therapy, or death from any cause, whichever occurs first.
Efficacy Endpoints 2:To evaluate the overall response rate after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Overall response rate (ORR), defined as the proportion of patients with a complete response (CR), complete response with incomplete bone marrow recovery (CRi), nodular partial response (nPR) or partial response (PR).
Efficacy Endpoints 3: To evaluate the duration of response after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Duration of response (DOR), defined as the time from the first documented response (PR or better) to disease progression or death (by any cause in the absence of disease progression).
Efficacy Endpoints 4: To evaluate the progression free survival after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Progression-free survival (PFS), defined as the time from randomisation to disease progression or death (by any cause in the absence of disease progression).
Efficacy Endpoints 5:To evaluate the event free survival after acalabrutinib treatment compared to investigators choice of treatment. | Visits are screening+ 8 visits( every 4 weeks) and then every 16 weeks until termination of the study which would be 4 years from the last subject randomized.
  Overall response rate (ORR), defined as the proportion of patients with a complete response (CR), complete response with incomplete bone marrow recovery (CRi), nodular partial response (nPR) or partial response (PR).

CONTACTS AND LOCATIONS:
Locations (22):
- United States (3):
  - Research Site, Charlotte, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
- Czechia (3):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Prague
- Italy (5):
  - Research Site, Cagliari
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Perugia
- Poland (2):
  - Research Site, Krakow
  - Research Site, Poznan
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
- United Kingdom (6):
  - Research Site, Bournemouth
  - Research Site, Oxford
  - Research Site, Plymouth
  - Research Site, Romford
  - Research Site, Stockton
  - Research Site, Sutton Coldfield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/